CLINICAL TRIAL: NCT03761251
Title: Pet Ownership and Glucose Control in Early Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Olga Gupta, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0044
Record Dates: First submitted 2018-11-28; First posted 2018-12-03 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 1; Adolescent Behavior
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pet Fish (Experimental): Participants will be instructed to partner thrice daily and once weekly fish care activities with diabetes care activities for 3 months
  Interventions: Behavioral: Pet Fish

INTERVENTIONS:
Behavioral: Pet Fish — Participants will be provided a fish tank with supplies to care for the fish and access to a fish (Betta splendens) from a local pet store. All participants will receive specific instructions for coupling the fish care and diabetes care:
  1. feed fish one pellet in the morning after waking; check and record BG reading at that time
  2. feed fish one pellet in the evening before dinner; check and record BG reading at that time
  3. feed fish one pellet at night before bedtime; check and record BG reading at that time
  4. every week clean the tank alternating with test the water quality in partnership with caregiver; review blood glucose readings with caregiver with each weekly fish care activity and problem solve any issues related to the blood glucose pattern.
  Each child will also receive two books intended to supplement and enrich their pet fish experience.

SUMMARY:
This study evaluates the short-term effects of incorporating the structured care of a pet fish into a diabetes self-care routine on glucose control in early adolescents with type 1 diabetes.

DETAILED DESCRIPTION:
Efficacy of treatment for Type 1 diabetes mellitus (T1DM) is dependent on adherence to self-care behaviors and collaborative parental involvement. Adolescence is a vulnerable time for the deterioration of glycemic control in patients with T1DM. In particular, parental monitoring declines during early adolescence. This often occurs before the child has developed self-efficacy and competence in independently performing diabetes-related tasks, including blood glucose monitoring. Consequently, there is a great need for innovative strategies in early adolescents that promote self-efficacy development and facilitate parental involvement.

ELIGIBILITY:
Inclusion Criteria:

* age 10-13 years
* diagnosis of T1DM
* duration of T1DM for at least one year
* fluency in English
* two recent consecutive HbA1c values 8.0 - 13%

Exclusion Criteria:

* clinical or laboratory characteristics suggestive of type 2 diabetes mellitus
* involvement in foster care
* dual-home living situation
* severe psychiatric disorders
* developmental delay or cognitive impairment
* current participation in another study that may impact glycemic control
* regular usage of a continuous glucose monitor
* HbA1c > 13% (because these individuals may need a more intensive intervention than this is intended to provide).

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 3 months
  Glycated hemoglobin test provides an average level of blood sugar over the past 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States